CLINICAL TRIAL: NCT01941368
Title: The Effects of β-Hydroxy-β-methylbutyrate Free Acid Gel and High-Intensity Interval Training on Quadriceps Muscle Architecture and Quality, Neuromuscular Economy, and Metabolic Performance in Recreationally Trained Individuals
Brief Title: The Effects of β-Hydroxy-β-methylbutyrate Free Acid and High-Intensity Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MTI2013-CS03; 13-257 (Other: University of Central Florida)
Record Dates: First submitted 2013-09-04; First posted 2013-09-13 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Exercise
Keywords: Performance; Aerobic Exercise
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Individuals assigned to Control Group will undergo baseline testing and then be asked to continue their normal exercise routine for 4 weeks and will undergo post-testing (visits 16 and 17) after this time period.
- Placebo + High-Intesnity Interval Training (HIIT) (Placebo Comparator): On training days, individuals will consume 1 gram of placebo 30 min prior to training, 1gram placebo 1 hour post training, and 1gram placebo 3 hours post training. On non-training days, individuals will consume placebo 3 times per day (8am, 12pm and 4pm).
  Interventions: Dietary Supplement: Placebo; Procedure: High Intensity Interval Training
- HMB-FA + HIIT (Active Comparator): On training days, individuals will consume 1 gram HMB-FA 30 min prior to training, 1gram HMB-FA 1 hour post training, and 1gram HMB-FA 3 hours post training. On non-training days, individuals will consume HMB-FA 3 times per day (8am, 12pm and 4pm).
  Interventions: Dietary Supplement: HMB-FA; Procedure: High Intensity Interval Training

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo + High-Intesnity Interval Training (HIIT)
Dietary Supplement: HMB-FA
  Other Names: beta-hydroxy-beta-methylbutyrate free acid (HMB-FA)
  Arms: HMB-FA + HIIT
Procedure: High Intensity Interval Training
  Arms: HMB-FA + HIIT; Placebo + High-Intesnity Interval Training (HIIT)

SUMMARY:
Objectives: 1) Determine the effect of 4-weeks of high intensity interval training (HIIT) and free acid form β-Hydroxy-β-methylbutyrate (HMB-FA) on VO2peak, lactate threshold, critical power, anaerobic working capacity and neuromuscular economy in a population of endurance trained individuals. 2) Determine the effect of 4-weeks of HIIT and HMB-FA on changes in skeletal muscle physiological cross-sectional area (PCSA=Volume/Fascicle length) and muscle quality (MQ=echo intensity) in the rectus femoris and vastus lateralis.

Subjects: Fifty males and females between the ages of 18 - 35 will be recruited to participate in this study. Subject will be randomized to one of three groups: a control group (CTL), an HIIT only group (HIIT) or a group which will take the amino acid metabolite HMB and perform HIIT (HMB-HIIT). Individuals assigned to CTL will undergo baseline testing. They will then be asked to continue their normal exercise routine for 4 weeks and will undergo post-testing after this time period.

Study Protocol: Two testing sessions, on nonconsecutive days, will occur at least 72 hours prior to the start of the training period. The same testing protocols will be repeated at the end of the 4-week training period. Testing protocols include performance testing (VO2peak, lactate threshold, critical power, anaerobic working capacity and neuromuscular economy) and anthropometric measures (physiological cross-sectional area and muscle quality). The training protocol for individuals in the experimental groups will consist of 4-weeks of high intensity interval training with three sessions per week on an electronically braked cycle ergometer. Individual work -loads will be calculated based on the outcomes from each participant's preliminary testing.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally-trained individuals with a VO2peak>40 ml∙kg-1∙min-1.
* Free of any physical limitations as determined by the Confidential Medical and Activity questionnaire and/or PAR-Q
* Between the ages of 18 and 35

Exclusion Criteria:

* Inability to perform physical exercise, as determined by the Confidential Medical and Activity questionnaire and/or PAR-Q
* Any chronic illness that causes continuous medical care

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
VO2peak/Ventilatory Threshold/fatigue threshold | Change from baseline after four weeks of high intensity interval training
  A continuous graded exercise test will be performed on an electronically-braked cycle ergometer to determine maximal oxygen consumption (VO2peak) and the peak power output (PPO) in watts (W) at VO2peak.

SECONDARY OUTCOMES:
EMG Activity Assessment | Change from baseline after four weeks of high intensity interval training
  To assess EMG activity, a bipolar surface electrode arrangement will be placed over the muscles of the quadriceps. The EMG signals will be expressed as root mean square (RMS) amplitude values. During the leg extensor trial, electromyography (EMG) root mean square (RMS) amplitude values will be recorded

OTHER OUTCOMES:
Ultrasonography | Change from baseline after four weeks of high intensity interval training
  Skeletal muscle images will be collected of the thigh muscles. These images will provide an ability to rate the quality of the leg muscles and determine the physiological cross-sectional area of the muscle
Three-minute Critical Power test | Change from baseline four weeks of high intensity interval training
  The participant will have 60 seconds of unloaded cycling at 90 rpm, followed by an all-out three-minute effort with resistance being set as a function of pedaling rate.
Maximal Isometric Strength | Change from baseline after four weeks of high intensity interval training
  To obtain the maximum isometric strength (kilograms) participants will be positioned in a BioDex S4 isometric dynamometer in a seated position. The participants will then be instructed to exert their maximum strength when trying to extend the knee and to produce the strength as fast as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Stout, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Sport and Exercise Science, Orlando, Florida, United States

REFERENCES:
- [Derived] Robinson EH 4th, Stout JR, Miramonti AA, Fukuda DH, Wang R, Townsend JR, Mangine GT, Fragala MS, Hoffman JR. High-intensity interval training and beta-hydroxy-beta-methylbutyric free acid improves aerobic power and metabolic thresholds. J Int Soc Sports Nutr. 2014 Apr 26;11:16. doi: 10.1186/1550-2783-11-16. eCollection 2014. PMID 24782684